CLINICAL TRIAL: NCT01104610
Title: Target Volume With a Pressure Controlled Ventilator in Obesity Hypoventilation Syndrome With Persistent Oxygen Desaturations With Continuous Positive Airway Pressure
Brief Title: Target Volume Mode Controlled Ventilator in Obesity Hypoventilation Syndrome
Acronym: OVO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped by the sponsor
Sponsor: Breas Medical S.A.R.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OVO-2009
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Obesity Hypoventilation Syndrome
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NIV-PSV without Target Volume (Active Comparator): Pressure Support Non Invasive Ventilation without Target Volume
  Interventions: Device: Breas Vivo 40
- NIV-PSV with Target Volume (Active Comparator): Non Invasive Pressure Support Ventilation with Target Volume set
  Interventions: Device: Breas Vivo 40
- NIV-CPAP (Active Comparator): Pressure Support Ventilation in CPAP mode
  Interventions: Device: Breas Vivo 40

INTERVENTIONS:
Device: Breas Vivo 40 — The Vivo 40 will be used either in CPAP mode, PSV mode without Target Volume or PSV mode with Target Volume
  Other Names: Breas Vivo 40 target volume

SUMMARY:
The purpose of this study is to investigate the evolution of daytime partial pressure of carbon dioxide in the blood (PaCO2) after 6 weeks of noninvasive ventilation-pressure support ventilation (NIV-PSV) with target volume versus continuous positive airway pressure (CPAP) alone versus NIV-PSV.

DETAILED DESCRIPTION:
Compare the efficacy between 3 ventilation modes (CPAP, PSV and PSV with Target Volume) on patients with obesity hypoventilation syndrome already treated with CPAP but with persistent desaturations.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 20 to 75 years old.
* Body mass index > 32 kg/m2
* Nocturnal oxygen desaturation 5 mn ≤ 88% under CPAP,
* PaCO2 > 5,9 kPa in diurnal, spontaneous ventilation

Exclusion Criteria:

* Patients with COPD and VEMS/FVC < 65%
* Patients with CHF and periodic breathing (Ejection Fraction <40%)
* Patients with a recent respiratory decompensation in the month preceding inclusion

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Evolution of daytime PaCO2 of NIV without target volume, with Target volume and with CPAP alone | 6 weeks

SECONDARY OUTCOMES:
Evolution in dyspnea scores (BDI/TDI and Simon Score) | 6 weeks
Evolution of subjective and objective sleepness (Osler) | 6 weeks
Cardiovascular parameters on Arterial strength (pulse velocity) and Endothelial function (Post ischemic test) | 6 weeks
Evolution of blood inflammation (IL6, TNFα et CRP) | 6 weeks
Evolution of insulin résistance | 6 weeks
Compliance (hours of treatment) | 6 weeks
Evolution of quality of ventilation (Leaks, asynchronism, others events) | 6 weeks
Sleep quality (PSG) between the 3 groups at 6 weeks | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pepin, prof, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - CHU, Grenoble
  - GH Pitié-Salpétrière - Service de pneumologie et réanimation, Paris